CLINICAL TRIAL: NCT02640924
Title: Proton Beam Radiotherapy Versus Switching Control Radiofrequency Ablation for Patients With Medium (>3, ≦5 cm) or Large (>5, ≦7cm) Treatment-naive Hepatocellular Carcinoma
Brief Title: Proton Radiotherapy Versus Radiofrequency Ablation for Patients With Medium or Large Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shi-Ming Lin, Director of Liver Research Unit, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103-1278A3
Record Dates: First submitted 2015-12-07; First posted 2015-12-29 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma; Proton therapy; Radiation therapy; Switching control radiofrequency ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proton radiotherapy (Experimental): Proton radiotherapy will be totally 66 cobalt gray equivalent (CGE) in 10 fractions and delivered once daily, 5 fractions per week, over 2 weeks for HCC more than 1 cm away from the alimentary tract.
  Interventions: Radiation: Proton radiotherapy
- Radiofrequency Ablation (Experimental): Multiple-electrode radiofrequency with switch-controller system (ME-SWC RFA) can create a large coagulation necrosis volume and successful treat HCC sized more than 3 cm, extending to 8.5 cm. ME-SWC RFA system uses up to 3 electrodes parallel insertion to inside of the tumors with an equilateral triangular confirmation before initiation of ablation. The distances between electrodes are about 1.5-2 cm, estimated by ultrasound measuring. The switching machine is set on the auto-mode, and all electrodes work alternately and switching each other automatically after impendence surge.
  Interventions: Procedure: Radiofrequency Ablation

INTERVENTIONS:
Radiation: Proton radiotherapy
  Arms: Proton radiotherapy
Procedure: Radiofrequency Ablation
  Arms: Radiofrequency Ablation

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most common cancers in Taiwan, where chronic viral hepatitis is common. Patients with HCC typically have impaired liver function because of virus- or alcohol- induced cirrhosis and viral hepatitis, and only approximately 20% of them are appropriate candidates for surgery. The 5-year overall survival for patients treated by surgery is approximately 30%-70%. For those not treated with surgery, liver function affected by an underlying liver disease has a strong influence on clinical outcomes, and complicates treatment strategies further than for other tumors. Maximal preservation of normal liver volume and function is an important consideration in the choice of treatment.

Proton beam has been applied to HCC treatment in Japan for longer than a decade, and several retrospective results showed excellent 3-5 years local control rate ranging from 85-95% and nearly no major complications. The investigators also retrospectively reviewed 75 index tumors sized 3.1-7.0cm in 70 patients receiving multiple-electrode radiofrequency ablation with switching controller (ME-SWC RFA) treatments in the period between 1 January 2009 and 31 December 2011 (Oral report in Taiwan Digestive Disease Week, October, 2012). Estimated 1-, 2-, and 3-year cumulative overall survival rates and local control rates were 94%, 85%, 81% and 89%, 83%, 67%, respectively.

Since ME-SWC RFA is the present one of standard modalities for non-surgery, moderate to larger (3-7 cm) HCC, and based on retrospective studies the local control rate of proton therapy was better than radiofrequency ablation, this prospective trial is aimed to compare the effects of these two modalities in 3-7 cm HCC patients who are not candidates for surgery or refuse surgery. This prospective study has high possibility to confirm the role of proton beam in HCC.

Along with the clinical trial, the investigators will also use next generation sequencing (NGS) to exam gene expression profile of tumor samples and find out candidate genes related to local control, intrahepatic control (treatment out-field control in liver), regional lymph node relapse, distant metastasis, and treatment response in HCC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed hepatocellular carcinoma or lesion with typical triphasic CT or MRI imaging features for HCC
* Single tumor and tumor size > 3cm, ≦7cm in diameter
* Patients are unsuitable for resection or unwilling to accept surgery.
* Age ≥20 years old
* Eastern Cooperative Oncology Group performance status score of 0 or 1
* Child-Pugh score ≦ 8
* Willing to sign informed consent regarding participation in this study

Exclusion Criteria:

* Patients have received any treatment for HCC before this study
* Pregnancy/breast feeding women
* Tumor adjacent to bowel <1cm
* Extrahepatic metastasis
* Extrahepatic invasion
* Portal or hepatic vein tumor invasion/thrombosis
* Uncontrolled ascites
* Glomerular filtration rate (GFR) < 30 ml/min*
* Platelet count < 50,000/L*
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 5 years
* Ongoing medically significant active infection.
* MRI incompatible devices
* * Baseline laboratories results must be within the protocol range prior to sign informed consent. Repeat lab tests are permitted to evaluate eligibility during the Screening Period.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Local control rate (treatment in-field control rate) | 3-year

SECONDARY OUTCOMES:
Overall survival rate | 3-year
Intrahepatic control rate | 3-year
Distant metastasis free survival rate | 3-year
Local control rate (treatment in-field control rate) | 5-year
Overall survival rate | 5-year
Intrahepatic control rate | 5-year
Distant metastasis free survival rate | 5-year
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3-year
Patient report outcome - quality of life as assessed by the functional assessment of cancer therapy - hepatobiliary (FACT-Hep) | 3-year
  The data will be collected 17 times from enrollment to the 36th month after treatment. Specific measurement points are: baseline, day 3, day 7, day 14, month 1, month 3, then every 3 months to the 36th month after treatment.
Patient report outcome - fatigue as assessed by the functional assessment of cancer therapy (FACT-F) | 3-year
  The data will be collected 17 times from enrollment to the 36th month after treatment. Specific measurement points are: baseline, day 3, day 7, day 14, month 1, month 3, then every 3 months to the 36th month after treatment.
Patient report outcome - pain as assessed by the brief pain inventory-short form (BPI-SF) | 3-year
  The data will be collected 17 times from enrollment to the 36th month after treatment. Specific measurement points are: baseline, day 3, day 7, day 14, month 1, month 3, then every 3 months to the 36th month after treatment.
Patient report outcome - symptom distress as assessed by the Memorial symptom assessment scale-short form (MSAS-SF) | 3-year
  The data will be collected 17 times from enrollment to the 36th month after treatment. Specific measurement points are: baseline, day 3, day 7, day 14, month 1, month 3, then every 3 months to the 36th month after treatment.
Patient report outcome - treatment satisfaction as assessed by the functional assessment of chronic illness therapy-treatment satisfaction-general (FACIT-TS-G) | 3-year
  The data will be collected 17 times from enrollment to the 36th month after treatment. Specific measurement points are: baseline, day 3, day 7, day 14, month 1, month 3, then every 3 months to the 36th month after treatment.
Patient report outcome - quality of life as assessed by the EQ-5D-3L | 3-year
  The data will be collected 17 times from enrollment to the 36th month after treatment. Specific measurement points are: baseline, day 3, day 7, day 14, month 1, month 3, then every 3 months to the 36th month after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Ming Lin, MD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Linkou, Taoyuan District, Taiwan

REFERENCES:
- [Background] Kan Z, Zheng H, Liu X, Li S, Barber TD, Gong Z, Gao H, Hao K, Willard MD, Xu J, Hauptschein R, Rejto PA, Fernandez J, Wang G, Zhang Q, Wang B, Chen R, Wang J, Lee NP, Zhou W, Lin Z, Peng Z, Yi K, Chen S, Li L, Fan X, Yang J, Ye R, Ju J, Wang K, Estrella H, Deng S, Wei P, Qiu M, Wulur IH, Liu J, Ehsani ME, Zhang C, Loboda A, Sung WK, Aggarwal A, Poon RT, Fan ST, Wang J, Hardwick J, Reinhard C, Dai H, Li Y, Luk JM, Mao M. Whole-genome sequencing identifies recurrent mutations in hepatocellular carcinoma. Genome Res. 2013 Sep;23(9):1422-33. doi: 10.1101/gr.154492.113. Epub 2013 Jun 20. PMID 23788652
- [Result] Mizumoto M, Okumura T, Hashimoto T, Fukuda K, Oshiro Y, Fukumitsu N, Abei M, Kawaguchi A, Hayashi Y, Ookawa A, Hashii H, Kanemoto A, Moritake T, Tohno E, Tsuboi K, Sakae T, Sakurai H. Proton beam therapy for hepatocellular carcinoma: a comparison of three treatment protocols. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):1039-45. doi: 10.1016/j.ijrobp.2010.07.015. Epub 2010 Oct 1. PMID 20888707
- [Result] Seror O, N'Kontchou G, Ibraheem M, Ajavon Y, Barrucand C, Ganne N, Coderc E, Trinchet JC, Beaugrand M, Sellier N. Large (>or=5.0-cm) HCCs: multipolar RF ablation with three internally cooled bipolar electrodes--initial experience in 26 patients. Radiology. 2008 Jul;248(1):288-96. doi: 10.1148/radiol.2481071101. Epub 2008 May 15. PMID 18483229
- [Result] Lee J, Lee JM, Yoon JH, Lee JY, Kim SH, Lee JE, Han JK, Choi BI. Percutaneous radiofrequency ablation with multiple electrodes for medium-sized hepatocellular carcinomas. Korean J Radiol. 2012 Jan-Feb;13(1):34-43. doi: 10.3348/kjr.2012.13.1.34. Epub 2011 Dec 23. PMID 22247634
- [Result] Lee JM, Han JK, Kim HC, Kim SH, Kim KW, Joo SM, Choi BI. Multiple-electrode radiofrequency ablation of in vivo porcine liver: comparative studies of consecutive monopolar, switching monopolar versus multipolar modes. Invest Radiol. 2007 Oct;42(10):676-83. doi: 10.1097/RLI.0b013e3180661aad. PMID 17984764